CLINICAL TRIAL: NCT04435639
Title: Can an Adjustable Compression Garment Replace Compression Bandaging in the Treatment of Patients With Breast Cancer Related Upper Limb Lymphoedema? A Pilot RCT Study
Brief Title: Using an Adjustable Compression Garment for Secondary Upper Limb Lymphoedema
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Researcher unable to continue.
Sponsor: Institute of Technology, Sligo (Other)
Collaborators: Sligo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITSligo SG
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Lymphedema of Upper Arm
Keywords: Breast cancer related lymphoedema.; Compression bandaging.
MeSH Terms: interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: Pilot Randomised Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor was blinded to treatment allocation. They evaluated participant's prior to treatment commencing and after treatment has been completed and compression garment/ compression bandaging has been removed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MLD + Adjustable Compression Sleeve. (Experimental): Manual lymph drainage + Adjustable Compression Sleeve.
  Interventions: Other: Manual lymph drainage.; Device: Adjustable Compression Sleeve
- MLD + Coban Compression Bandage. (Active Comparator): Manual lymphatic drainage + Coban compression bandaging.
  Interventions: Other: Manual lymph drainage.; Procedure: Coban compression bandage..

INTERVENTIONS:
Other: Manual lymph drainage. — Manual Lymphatic drainage:
  Patients will receive manual lymphatic drainage by massage for 40 minutes for 5 treatments over a 15 day period.
Procedure: Coban compression bandage.. — Coban compression bandaging: Patients will be wrapped in Coban compression bandaging which stays on until the next treatment. Patients will wear standard compression sleeves during the six month maintenance phase.
  Arms: MLD + Coban Compression Bandage.
Device: Adjustable Compression Sleeve — Patients wear an adjustable compression sleeve (Juzo varocare adjustable compression system) between treatments. They will be shown how to put it on and how to tighten the sleeve when needed. Patients will also wear the adjustable compression sleeve in alternation with a standard compression sleeve over a six month maintenance phase.
  Arms: MLD + Adjustable Compression Sleeve.

SUMMARY:
This is a pilot randomised controlled trial investigating the use of an adjustable compression garment in the treatment of patients with Breast Cancer related upper limb Lymphoedema. This study will be conducted as part of a MSc qualification at the Institute of Technology Sligo in Ireland with all therapy sessions taking place in the Physiotherapy Department of Sligo University Hospital (formerly Sligo General Hospital). The study will be conducted in conjunction with Sligo University Hospital and it has attained ethical approval through the relevant University Hospital Ethics Committee.

DETAILED DESCRIPTION:
The experimental group will receive 5 treatments followed by a final assessment on the 6th visit over a 3 week period: participants will receive manual lymphatic drainage for 40 minutes. They will then put on an Adjustable Compression sleeve (Juzo varocare adjustable compression system). Patients will be re-measured before the fourth treatment and again on session 6. At this point patients will receive a standard arm compression sleeve. This will be worn in alternation with their adjustable compression sleeve over the following 6 months. Patient will have their limb volume re-measured at the 6 month review.

The control group will receive 5 treatments followed by a final assessment on the 6th visit over a 3 week period: participants will receive manual lymphatic drainage for 40 minutes. They will then have their arm wrapped in Coban compression bandaging which will stay on until their next treatment. This will occur twice weekly for a period of 3 weeks. Patients will be Re-measured before the fourth treatment and again on session 6. At this point they will attend occupational therapy where they will receive 2 standard arm compression sleeves. The patient wears 1 sleeve every day over the following 6 months. Patient will have their limb volume re-measured at the 6 month review.

ELIGIBILITY:
Inclusion Criteria:

* Upper limb lymphoedema (secondary to breast cancer) diagnosed by a consultant
* Aged > 18 years.
* Males and females.
* Stage 2 Lymphoedema.
* >10% volume difference between upper limbs.
* Cognitive ability to understand the programme.

Exclusion Criteria:

* Involvement in other studies or rehabilitation programmes.
* Active infection disease progression.
* Congestive Cardiac Failure.
* Non-English speakers.
* Under 18's.
* Poor cognition for treatment compliance or consent.
* Pregnant, or currently breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Limb Volume - Circumferential Measurements. | Over a 6 month period. (10 min testing time)
  Limb Volume- circumferential measurements taken at 4cm intervals from the wrist up to the axilla.
  The circumferences were then entered into a spreadsheet and a truncated cone formula applied with each segment volume calculated: Vs = h(Ct x Ct + Ct x Cb x Cb) 12 π
  where (Vs) was volume of a segment, (h) was the distance between two points of measurement, (Ct) represented the circumference at the top measurements of the segment, (Cb) represented the circumference at the base of the segment, π = Pi. Once each segment is calculated, the sum of all segments of the arm are computed into a volume estimate. This method was found to be valid (criterion validity)in several studies when compared to the gold standard of water displacement with intra-class correlation coefficient (ICC) of >0.95. The higher the score the more lymphoedema present.
Short Form 36 (SF-36): Quality of Life questionnaire. | Over a 6 month period. (10 min testing time)
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting for routine monitoring and assessment of care outcomes in adult patients.It is scored 0-100 with a lower score indicating more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Shane Gallagher, MSc, Principal Investigator — Study Principal Investigator
Locations (1):
- Atlantic Technological University, Sligo, Ireland

DOCUMENTS (3):
  • Study Protocol (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT04435639/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT04435639/SAP_001.pdf
  • Informed Consent Form (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT04435639/ICF_002.pdf